CLINICAL TRIAL: NCT07047885
Title: A Phase I/IB Study of Ropeginterferon in Patients With Cutaneous T-Cell Lymphoma (CTCL)
Brief Title: Ropeginterferon in Patients w/Cutaneous T-Cell Lymphoma (CTCL)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: PharmaEssentia (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MCC-23455
Record Dates: First submitted 2025-06-23; First posted 2025-07-02 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Cutaneous T Cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dose Level -2 (Experimental): 250 µg SQ every 2 weeks
  Interventions: Drug: Ropeginterferon alfa-2b
- Dose Level -1 (Experimental): 350 µg SQ every 2 weeks
  Interventions: Drug: Ropeginterferon alfa-2b
- Dose Level 1 (Experimental): 500 µg SQ every 2 weeks
  Interventions: Drug: Ropeginterferon alfa-2b
- Expansion Arm (Experimental): Once the Recommended Phase 2 Dose (RP2D) is reached, an additional 20 participants will be treated at this dose for additional experience with safety and efficacy.
  Interventions: Drug: Ropeginterferon alfa-2b

INTERVENTIONS:
Drug: Ropeginterferon alfa-2b — Will be administered via subcutaneous injection once every 2 weeks
  Other Names: P1101

SUMMARY:
This is a single-center, phase I/IB study to identify the recommended phase II dose of Ropeginterferon-alfa 2b (P1101) in patients with CTCL who have failed at least two prior lines of skin-directed therapy (Stage IA-IB) or have less than a complete response to phototherapy or extracorporeal photopheresis (ECP) or total skin electron beam therapy (TSET), or stable/progressive disease after at least two lines of topical therapy (Stage IIA-IIIB).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with cutaneous T-cell lymphoma, stage IA-IIIB CTCL according to WHO-EORTC classification, specifically the following subtypes: Mycosis Fungoides (MF); Sézary Syndrome (SS); Lymphomatoid Papulosis (LyP) or other rare CTCL variants per WHO-EORTC classification, provided the investigator determines the disease course warrants systemic treatment.
* A) For Stage IA-IB: Must have failed at least two prior lines of skin-directed therapy, where "failed" is defined as any of the following: a. Inadequate response (persistent clinically significant lesions or symptoms), b. Unacceptable toxicity, or c. Disease progression. Such patients require a systemic approach because of symptomatic, refractory, or recalcitrant disease. B) For Stage IIA-IIIB: Must have a documented less-than-complete response to phototherapy, extracorporeal photopheresis (ECP), or total skin electron beam therapy (TSET), or have failed disease after ≥2 lines of topical therapy (using the same definition of "failed" as above.
* Patients are allowed to continue phototherapy or ECP at their prior schedule or a less frequent schedule. Topical therapy, phototherapy, and ECP are allowed if the patient has been on a stable dose of topical therapy or schedule of the phototherapy or ECP. Patients are not allowed to start new skin-directed therapies or escalate the frequency of the prior skin-directed therapy schedule while on the study.
* Male or female, aged 18 years or older.
* There is no evidence of large cell transformation on the skin biopsy at the screening visit.
* Ability to take subcutaneous injection medication and be willing to adhere to the P1101 q2week injection regimen.
* Minimum wash-out period of 3 weeks between the last dose of prior systemic therapy (other anti-cancer therapy aside from ECP or phototherapy) and the first dose of P1101.
* Women of childbearing potential (WCBP) must have a negative serum beta-HCG pregnancy test within 7 days of receiving study medication. An WOCP is considered a sexually mature female who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 12 consecutive months. For WOCP and female partners of male subjects, reliable contraception methods must be used throughout the duration of treatment up to at least 8 weeks after the last dose of study drug has been administered.
* Ability to understand and the willingness to sign a written informed consent document.
* Acceptable Hematologic Parameters
* Thyroid-stimulating hormone (TSH) within institutional normal limits OR well-controlled on thyroid replacement.
* Lipid Panel: a. No severe hypertriglyceridemia (e.g., triglycerides < 400-500 mg/dL, or medically manageable per investigator discretion). b. No uncontrolled hypercholesterolemia that is unresponsive to standard lipid lowering agents.
* Renal Function: Estimated glomerular filtration rate (eGFR) ≥ 30 mL/min using a CKD EPI.
* AST/ALT < 3 x upper limit of normal (ULN), and total bilirubin < 2 x ULN (unless due to Gilbert's syndrome).

Exclusion Criteria:

* Large cell transformation at screening visit.
* Child-Pugh B or C hepatic impairment of any etiology.
* Uncontrolled psychiatric disorders, defined as Patient Health Questionnaire-2 (PHQ-2) depression screening score equal to or above 3.
* Treatment with another investigational drug or other systemic drug within 3 weeks. Concomitant administration of radiotherapy or systemic anti-cancer therapy, including but not restricted to chemotherapy, biological agents, or immunotherapy. Concurrent use of systemic steroids is allowed in patients with erythroderma who have been on corticosteroids to avoid possible rebound flare of the disease, adrenal insufficiency, or unnecessary suffering. Concomitant phototherapy or extracorporeal photopheresis (ECP) are also allowed.
* Severe or unstable cardiovascular disease (uncontrolled hypertension, heart failure (≥ NYHA class 2), serious cardiac arrhythmia, significant coronary artery stenosis, unstable angina, or recent stroke or myocardial infarction.
* Active, uncontrolled HIV, detectable HBV, or active HCV infection. The patients who are stable on anti-retroviral therapy or suppressed on HBV/HCV therapy are allowed in the study.
* Active, uncontrolled ophthalmic disorders such as severe retinopathy, uncontrolled glaucoma, or advanced proliferative retinopathy.
* History of or active serious or uncontrolled autoimmune disease, or patients on systemic immunosuppressants or history of systemic immunosuppressants for autoimmune disease.
* History of solid organ or stem cell transplantation recipients who are at heightened risk for immunologic complications on interferons.
* Known hypersensitivity to interferons.
* Baseline QTcF > 470 ms.
* No active, serious infection requiring systemic antimicrobial therapy at screening.
* Pregnant or breastfeeding women are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2025-08-27 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity | 6 weeks
  The percentage of participants who experience any grade 3 or higher non-hematologic toxicity and grade 4 or higher hematologic toxicity of P1101 according to CTCAE v5.0 during the first six weeks of therapy.
Recommended Phase II Dose | 6 weeks
  The Recommended Phase II Dose will be determined according to the Bayesian optimal interval (BOIN) design.

SECONDARY OUTCOMES:
Overall Response Rate | 1 year
  Proportion of patients who achieve a complete response or a partial response.

CONTACTS AND LOCATIONS:
Overall Officials: Yumeng Zhang, MD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States